CLINICAL TRIAL: NCT05346744
Title: Quantitative Clinical Evaluation of the Occlusal Contact Trueness Affected by Six Chairside CAD/CAM Ceramic Materials：a Self-control Study
Brief Title: Occlusal Contact Trueness Affected by Six Chairside CAD/CAM Ceramic Materials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Hao Yu, vice dean of school and hospital of stomatology, Fujian Medical University
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2019028
Record Dates: First submitted 2022-04-15; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Tooth Defect
Keywords: chairside CAD/CAM; ceramic materials; trueness; occlusal contact

STUDY DESIGN:
Intervention Model Description: Ten individuals with tooth defect of mandibular first molar were selected to participate in the study. 6 crowns made from 6 chairside materials were milled by CEREC MCXL-EF mode for each mandibular first molar.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Care providers and outcomes assessors wouldn't know the materials of the specimen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Zirconia (Experimental): 10 crowns made of zirconia from 10 individual were milled, post-processed and occlusal adjusted in patients' mouth.
  Interventions: Other: Chairside CAD/CAM ceramic materials for dental restoration
- Celtra Duo (Experimental): 10 crowns made of Celtra Duo from 10 individual were milled, post-processed and occlusal adjusted in patients' mouth.
  Interventions: Other: Chairside CAD/CAM ceramic materials for dental restoration
- e.max CAD (Experimental): 10 crowns made of e.max CAD from 10 individual were milled, post-processed and occlusal adjusted in patients' mouth.
  Interventions: Other: Chairside CAD/CAM ceramic materials for dental restoration
- Lici UPCERA (Experimental): 10 crowns made of Lici from 10 individual were milled, post-processed and occlusal adjusted in patients' mouth.
  Interventions: Other: Chairside CAD/CAM ceramic materials for dental restoration
- Enamic (Experimental): 10 crowns made of Enamic from 10 individual were milled, post-processed and occlusal adjusted in patients' mouth.
  Interventions: Other: Chairside CAD/CAM ceramic materials for dental restoration
- Runci UPCERA (Experimental): 10 crowns made of Runci from 10 individual were milled, post-processed and occlusal adjusted in patients' mouth.
  Interventions: Other: Chairside CAD/CAM ceramic materials for dental restoration

INTERVENTIONS:
Other: Chairside CAD/CAM ceramic materials for dental restoration — 6 crowns made from 6 chairside ceramic materials were milled by CEREC MCXL-EF mode for mandibular first molar of each participant.
  The six materials are as follows:
  ZIR: InCoris TZI (Dentsply Sirona, York, PA)， CD: Celtra Duo (Dentsply Sirona, York, PA), EMA: e.max CAD (ivoclar, Vivadent AG), LC: LiCi (UPCERA, China), ENA: Vita Enamic (Vita Zahnfabrik, Bad Sackingen, Germany) RC: RunCi (UPCERA, China)

SUMMARY:
The aim of this clinic self-control study was to evaluate the trueness of occlusal contact affected by six ceramic materials during chairside fabricating process and offer recommendations for occlusal offset according to different ceramic materials in CEREC CAD/CAM design process.

DETAILED DESCRIPTION:
Ten participants were selected for this study. InCoris TZl(ZIR), Celtra Duo(CD), IPS e.max(EMA), UPCERA LICI (LC), Vita enamic(ENA), UPCERA RUNCI (RC) were used to produce crowns for everyone by CEREC chairside CAD/CAM system. The milling trueness, postprocessing trueness and clinical adjustment of occlusal contact were quantitatively analyzed by the ATOS high-precision scanner and Geomagic reverse engineering software.

ELIGIBILITY:
Inclusion Criteria:

1. with one mandibular first molar requiring crown restoration that have undergone root canal treatment;
2. with complete permanent dentition;

Exclusion Criteria:

1. with carious lesions, abrasions, attrition, erosions or any kind of tooth defects;
2. with any kind of restorations in occlusal surfaces;
3. with any sign of temporomandibular dysfunction.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
milling trueness(μm) | 1 week
  the absolute 3D deviation of occlusal contact points before and after milling
postprocessing trueness(μm) | 1 week
  the absolute 3D deviation of occlusal contact points before and after postprocessing
clinical trueness(μm) | 1 week
  the absolute 3D deviation of occlusal contact points before and after occlusal adjustment

CONTACTS AND LOCATIONS:
Overall Officials: Hao Yu, Principal Investigator — Fujian Medical University
Locations (1):
- Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT05346744/Prot_SAP_000.pdf